CLINICAL TRIAL: NCT05731388
Title: Assessing Depth of Small Bowel Insertion at Push Enteroscopy by Using Capsule Endoscopy to Determine Best Diagnostic Approach for Patients With Obscure Gastrointestinal Bleeding
Brief Title: Assessing Depth of Small Bowel Insertion at Push Enteroscopy by Using Capsule Endoscopy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 19-037
Record Dates: First submitted 2022-10-28; First posted 2023-02-16 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Obscure Gastrointestinal Bleeding; Gastrointestinal Diseases; Gastrointestinal Bleed; Angiodysplasia Intestine
MeSH Terms: conditions — Gastrointestinal Diseases; Gastrointestinal Hemorrhage | interventions — Double-Balloon Enteroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Push enteroscopy — A push enteroscopy using a pediatric colonoscope will be performed along with capsule endoscopy. These are part of the standard of care.

SUMMARY:
Bleeding from the gastrointestinal tract can originate from the small bowel. Typically, upper and lower endoscopies are unable to identify the site of bleeding and patients need to undergo special endoscopies with longer cameras to examine the small bowel and find the bleeding site. One of the most commonly used scopes to investigate the first part of the small intestinal is called "push enteroscopy". This is an upper endoscopy that uses a pediatric colonoscope, which is longer. To date, it is unknown what percentage of small bowel can be observed with this technique. Hence, this study aimed to determine the extent of small bowel examined by push enteroscopy. Consecutive patients with suspected bleeding from the small intestine will undergo a push enteroscopy and the depth of the examination will be marked with metallic clips. Subsequently, patients will have a capsule endoscopy, which is a little camera that will take multiple pictures of the whole small intestine. The percentage of small bowel that the push enteroscopy examined will be determined by the percentage of small bowel corresponding to the location of the clips visualized on capsule endoscopy.

DETAILED DESCRIPTION:
Consecutive adult patients (aged > 18 years) referred to a single tertiary referral center for investigation of OGIB will be prospectively recruited. Patients will be included if they had overt signs of GI bleeding (hematochezia or melena with an associated drop in hemoglobin) or occult signs of GI bleeding in the form of persistent or recurrent iron deficiency anemia and had undergone esophagogastroduodenoscopy (EGD) and colonoscopy that were negative for a source of bleeding. Exclusion criteria include significant cardiopulmonary disease, an implanted electromedical device, pregnancy, previous gastrectomy, extensive Crohn's disease with suspicion for stricturing or fistulizing small bowel disease. All patients will provide informed consent before enrollment.

The study protocol was approved by the Institutional Review Board (IRB) at our institution and was conducted in accordance with ethical guidelines of the Helsinki Declaration Procedures Patients will undergo bowel preparation by oral ingestion of 2L of polyethylene glycol solution 12 hours before the study. Push enteroscopy (PE) will be performed in an endoscopy theater with patients under conscious sedation using intravenous injections of midazolam (0.05-0.1mg/kg) and fentanyl (1-2 mcg/kg), with dimenhydrinate (25-50mg/body) added in the case of insufficient sedation. Cardiorespiratory function will be monitored during the procedure. Antiplatelet and anticoagulant medications will be discontinued 3-7 days before the procedure. No intravenous antispasmodic will be used during the PE in efforts to preserve normal gut motility for the passage of the subsequent capsule endoscopy (CE). A pediatric colonoscope furnished with a water-jet system (PCF-TYPE H190L; Olympus Co, Tokyo, Japan) and distal transparent attachment cap will be inserted through the mouth and be advanced as far as possible into the small bowel using a water immersion technique and aided by multiple reduction maneuvers. No overtube will be used and carbon dioxide will be used for insufflation in all cases. Two endoscopic clips (SureClip; Micro-Tech Co, Nanjin, China) will be placed at the maximal distal insertion point to mark this location for identification by CE. The endoscope will be then withdrawn gradually as per our standard practice for direct examination of the small bowel traversed by the PE. The presence of any vascular or non-vascular lesions will be recorded and endoscopic treatments such as argon plasma coagulation (APC), endoscopic clips or biopsies will be performed as clinically appropriate depending on the nature of the lesions found. In particular, the number of vascular lesions seen and how many of these lesions were treated with APC will be recorded. After PE is completed, the capsule (PillCam TM SB3 capsule; Medtronic, Dublin, Ireland) synchronized with the recording device will be deployed into the first part of the duodenum by using a gastroscope (GIF-HQ190; Olympus, Tokyo, Japan) and capsule deployment device (AdvanCE Endoscope Delivery Device; STERIS, OH, USA). Capsule recording devices will be retrieved 8-12 hours after capsule deployment and images read by two separate endoscopists trained in reporting CE. CE recordings will be reviewed using the RAPID 8.0 software. The location of the clip placed at the deepest insertion point of the PE as seen by CE will be quantified by the percentage of small bowel progress (SBP) and small bowel transit time (SBTT) from the duodenal bulb to the clip relative to the entire length of the small intestine from the duodenal bulb to the cecum. Any bleeding lesions and their respective locations will also be recorded. Furthermore, the number of angioectasias treated during PE that were seen again on CE will be recorded to calculate the detection rates of these lesions.

The primary outcome of the study is to estimate the proportion of the small intestine that can be evaluated by using the PE technique. Secondary outcomes include the diagnostic yield of CE and PE in identifying the cause of obscure gastrointestinal bleeding, comparison of the detection rates between the two modalities and adverse events related to these procedures. Statistical analyses will be performed using JMP Pro 15 (SAS Institute, Cary, NC, USA). Continuous variables will be expressed as a mean with standard deviation (SD) or 95% confidence interval (CI), or median with interquartile range (IQR) according to distribution.

ELIGIBILITY:
Inclusion Criteria:

* Patients with overt signs of GI bleeding (OGIB) (hematochezia or melena with an associated drop in hemoglobin) or occult signs of GI bleeding in the form of persistent or recurrent iron deficiency anemia and had undergone esophagogastroduodenoscopy (EGD) and colonoscopy that were negative for a source of bleeding.

Exclusion Criteria:

* Significant cardiopulmonary disease, an implanted electromedical device, pregnancy, previous gastrectomy, extensive Crohn's disease with suspicion for stricturing or fistulizing small bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients (aged > 18 years) referred to a single tertiary referral center for investigation of OGIB will be prospectively recruited
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of small bowel examination | through study completion, an average of 3 years
  Proportion of the small intestine that can be evaluated by using the PE technique.

SECONDARY OUTCOMES:
Diagnostic yield of CE and PE in identifying the cause of obscure gastrointestinal bleeding, comparison of the detection rates between the two modalities and adverse events related to these procedures | through study completion, an average of 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Teshima, MD MSc PhD, Principal Investigator — Unity Health Toronto, St. Michael's Hospital
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barkin JS, Lewis BS, Reiner DK, Waye JD, Goldberg RI, Phillips RS. Diagnostic and therapeutic jejunoscopy with a new, longer enteroscope. Gastrointest Endosc. 1992 Jan-Feb;38(1):55-8. doi: 10.1016/s0016-5107(92)70333-2. No abstract available. PMID 1612382
- [Background] Cortegoso Valdivia P, Skonieczna-Zydecka K, Pennazio M, Rondonotti E, Marlicz W, Toth E, Koulaouzidis A. Capsule endoscopy transit-related indicators in choosing the insertion route for double-balloon enteroscopy: a systematic review. Endosc Int Open. 2021 Feb;9(2):E163-E170. doi: 10.1055/a-1319-1452. Epub 2021 Jan 25. PMID 33532554